CLINICAL TRIAL: NCT02963649
Title: Randomized Study of IN.PACT 014 Paclitaxel-Coated Percutaneous Transluminal Angioplasty Balloon Catheter vs. Optimal Percutaneous Transluminal Angioplasty for the Treatment of Chronic Total Occlusions in the Infrapopliteal Arteries
Brief Title: IN.PACT BTK Randomized Study to Assess Safety and Efficacy of IN.PACT 014 vs. PTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APV-IN.PACT BTK OUS
Record Dates: First submitted 2016-11-09; First posted 2016-11-15 (Estimated); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Coated Balloon IN.PACT 014 (DCB) (Experimental): Participants who receive IN.PACT 014.
  Interventions: Device: DCB
- Percutaneous Transluminal Angioplasty (PTA) (Active Comparator): Participants who receive standard PTA treatment.
  Interventions: Device: PTA

INTERVENTIONS:
Device: DCB — Drug Coated Balloon
  Arms: Drug Coated Balloon IN.PACT 014 (DCB)
Device: PTA — Percutaneous Transluminal Angioplasty
  Arms: Percutaneous Transluminal Angioplasty (PTA)

SUMMARY:
To assess the safety and efficacy of the paclitaxel drug-coated balloon IN.PACT 014 versus conventional optimal percutaneous transluminal angioplasty (PTA) for the treatment of patients with chronic total occlusions in the infrapopliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Subject has been informed of the nature of the study, agrees to participate and has signed an EC approved consent form.
3. Female subjects of childbearing potential have a negative pregnancy test ≤7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation.
4. Subject has documented chronic Critical Limb Ischemia (CLI) in the target limb prior to the study procedure with Rutherford Clinical Category 4 or 5.
5. Subjects with documented infection grade 0-2 and ischemia grade 2-3 according to WIfi classification.
6. Life expectancy >1 year in the Investigator's opinion.
7. Reference Vessel Diameter (RVD) 2 - 4 mm, and confirmed by DUS assessment.
8. Total occlusions with total lesion length ≥ 40 mm (by visual estimate).
9. Lesion must be located in the infrapopliteal arteries and above the ankle joint.
10. Multiple lesions can be treated if located in separate vessels.
11. Presence of documented run-off to the foot.
12. Inflow free from flow-limiting lesion confirmed by angiography.
13. Successful pre-dilatation of the (entire) target lesion.

Exclusion Criteria:

1. Subject unwilling or unlikely to comply to the appropriate follow-up times for the duration of the study.
2. Planned index limb amputation above the metatarsal level, or any other planned major surgery within 30 days pre or post-procedure.
3. Lesion and/or occlusions located or extending in the popliteal artery or below the ankle joint space.
4. Significant (≥50% DS) inflow lesion or occlusion in the ipsilateral iliac, SFA and popliteal arteries left untreated.
5. Failure to obtain ≤ 30% residual stenosis in pre-existing, hemodynamically significant inflow lesions in the ipsilateral iliac, SFA and popliteal artery.
6. Prior stent(s) or bypass surgery within the target vessel(s) (including stents placed within target vessels during the index procedure prior to randomization.
7. Previous DCB procedure in the target vessel within 6 months prior to index procedure.
8. Aneurysm in the target vessel.
9. Angiographic evidence of thrombus within target limb.
10. Pre-dilatation resulted in major (≥ Grade D) flow-limiting dissection or residual stenosis > 30%.
11. Use of alternative therapy e.g. atherectomy, cutting balloon, laser, radiation therapy, stents as part of target vessel treatment.
12. Recent MI or stroke < 30 days prior to the index procedure.
13. Heart failure with Ejection Fraction < 30%.
14. Known or suspected active infection at the time of the index procedure, excluding an infection of a lower extremity wound on the target limb.
15. Subjects with infection grade 3 and ischemia grade 0 and 1 according to the Wifi classification.
16. Subjects with neutrotrophic ulcers, heel pressure ulcers or calcaneal ulcers with a risk of major amputation.
17. Subjects with documented active osteomyelitis, excluding the phalanges, that is beyond cortical involvement of the bone per clinical judgement.
18. Impaired renal function (GFR <20 mL/min) and patients on dialysis.
19. Subject with vasculitis, systemic Lupus Erythematosus or Polymyalgia Rheumatica on active treatment.
20. Patient receiving systemic corticosteroid therapy.
21. Known allergies or sensitivities to heparin, aspirin (ASA), other anticoagulant/anti-platelet therapies which could not be substituted, and/or paclitaxel or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.
22. The patient is currently enrolled in another investigational device or drug trial that is interfering with the endpoints of this study.
23. Female subjects who are breastfeeding at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Belgium (3):
  - AZ Sint Blasius, Dendermonde, East-Flanders
  - ZOL Genk, Genk, Limburg
  - Universitair Ziekenhuis Gent, Ghent
- Hopital Guillaume et Rene Laennec - Centre Hospitalier Universitaire, Nantes, France
- University Hospital Patras, Pátrai, Greece
- Italy (3):
  - IRCCS Multimedica, Sesto San Giovanni, Lombardy
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - Ospedale San Donato, Arezzo
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liistro F, Weinberg I, Almonacid Popma A, Shishehbor MH, Deckers S, Micari A. Paclitaxel-coated balloons versus percutaneous transluminal angioplasty for infrapopliteal chronic total occlusions: the IN.PACT BTK randomised trial. EuroIntervention. 2022 Apr 1;17(17):e1445-e1454. doi: 10.4244/EIJ-D-21-00444. PMID 34602386

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug Coated Balloon IN.PACT 014: Participants who receive IN.PACT 014
Period: Overall Study
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Started | 23 (23 Participants were enrolled in the IN.PACT 014 arm. For Primary and Secondary Outcome measures, the Overall Number of Participants Analyzed may differ from the number reported in the row in the Participant Flow module, due to missing data for the respective Outcome measure.) | 27 (27 Participants were enrolled in the PTA arm. For Primary and Secondary Outcome measures, the Overall Number of Participants Analyzed may differ from the number reported in the row in the Participant Flow module, due to missing data for the respective Outcome measure.)
Completed | 11 | 16
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Population: Study sites identified 25 target lesions in the IN.PACT 014 group and 30 in the PTA group. All site-reported lesion characteristics use 25 as the denominator for the IN.PACT 014 group and 30 as the denominator for the PTA group. CoreLab identified 24 target lesions in the IN.PACT 014 group and 29 in the PTA group. Therefore, all CoreLab reported lesion characteristics use 24 as the denominator for the IN.PACT 014 group and 29 as the denominator for the PTA group.
Units Other Than Participants: Lesions
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA) | Total
Number analyzed (Participants) | 23 | 27 | 50
Number analyzed (Lesions) | 25 | 30 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.1 (7.4) | 69.6 (9.4) | 71.20 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 19 | 20 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Obesity, BMI >=30kg/m2 [Count of Participants; unit: Participants] — Population: Denominator is subjects with available data.
  Participants
    number analyzed (Participants) | 22 | 26 | 48
    (all) | 5 | 7 | 12
Diabetes Mellitus [Count of Participants; unit: Participants] | 17 | 26 | 43
Diabetes Mellitus Insulin-dependent [Count of Participants; unit: Participants] | 9 | 20 | 29
Hypertension [Count of Participants; unit: Participants] | 19 | 21 | 40
Hyperlipideamia [Count of Participants; unit: Participants] — Population: Denominator is subjects with available data.
  Participants
    number analyzed (Participants) | 22 | 25 | 47
    (all) | 16 | 20 | 36
Current smoker [Count of Participants; unit: Participants] — Population: Denominator is subjects with available data.
  Participants
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 4 | 3 | 7
End-stage renal disease [Count of Participants; unit: Participants] | 0 | 0 | 0
Cerebrovascular disease [Count of Participants; unit: Participants] — Population: Denominator is subjects with available data.
  Participants
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 6 | 3 | 9
Congestive heart failure [Count of Participants; unit: Participants] — Population: Denominator is subjects with available data.
  Participants
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 2 | 5 | 7
Ischaemic heart disease [Count of Participants; unit: Participants] — Population: Denominator is subjects with available data.
  Participants
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 10 | 9 | 19
Bilateral PAD [Count of Participants; unit: Participants] — Population: Denominator is subjects with available data.
  Participants
    number analyzed (Participants) | 22 | 22 | 44
    (all) | 12 | 14 | 26
Previous peripheral revascularisation of target limb [Count of Participants; unit: Participants] | 7 | 9 | 16
Previous minor target limb amputation [Count of Participants; unit: Participants] | 3 | 11 | 14
Rutherford category 4 [Count of Participants; unit: Participants] — RUTHERFORD-BECKER SCALE (Clinical Category) 4 = Ischemic rest pain. Increased score is a worse outcome for Critical Limb Ischemia.
  Participants | 3 | 3 | 6
Rutherford category 5 [Count of Participants; unit: Participants] — RUTHERFORD-BECKER SCALE (Clinical Category) 5 = Minor tissue loss, focal gangrene with diffuse pedal ischemia.
  Increased score is a worse outcome for Critical Limb Ischemia.
  Participants | 20 | 24 | 44
Rutherford category 6 [Count of Participants; unit: Participants] — RUTHERFORD-BECKER SCALE (Clinical Category) 6 = Major tissue loss-extending transmetatarsally; functional foot no longer salvageable.
  Increased score is a worse outcome for Critical Limb Ischemia.
  Participants | 0 | 0 | 0
Target lesion location - Popliteal P3 segment [Count of Units; unit: Lesions] — Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 2 | 1 | 3
Target lesion location - Tibio-peroneal trunk [Count of Units; unit: Lesions] — Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 4 | 4 | 8
Target lesion location - Anterior tibial [Count of Units; unit: Lesions] — Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 17 | 15 | 32
Target lesion location - posterior tibial [Count of Units; unit: Lesions] — Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 6 | 12 | 18
Target lesion location - Peroneal [Count of Units; unit: Lesions] — Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 1 | 2 | 3
Inflow in the target vessel (<30% residual stenosis) [Count of Participants; unit: Participants] — Population: Participant-based assessment. Denominator is subjects with available data.
  Participants
    number analyzed (Participants) | 20 | 24 | 44
    (all) | 18 | 21 | 39
Lesion type - De novo [Count of Units; unit: Lesions] — Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement. Number of Participants DCB = 23; Number of Participants PTA = 27; Total Number of Participants = 50.
  Lesions | 20 | 26 | 46
Lesion type - Restenotic (non-stented) [Count of Units; unit: Lesions] — Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement. Number of Participants DCB = 23; Number of Participants PTA = 27; Total Number of Participants = 50.
  Lesions | 5 | 4 | 9
Lesion length [Mean (Standard Deviation); unit: mm] — Population: Lesion based measurement. CoreLab reported data; Overall N Lesions DCB = 24; Overall N Lesions PTA = 29
  Participant analysis not performed, as this is a lesion-based measurement.
  mm
    number analyzed (Participants) | 23 | 26 | 49
    number analyzed (Lesions) | 24 | 28 | 52
    (all) | 215.41 (83.81) | 218.19 (80.43) | 216.91 (81.20)
Occluded lesion (site reported data) [Count of Units; unit: Lesions] — Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement. Number of Participants DCB = 23; Number of Participants PTA = 27; Total Number of Participants = 50.
  Lesions | 25 | 30 | 55
Total occluded lesion length, mm [Mean (Standard Deviation); unit: mm] — Population: Lesion based measurement. CoreLab reported data; Overall N Lesions DCB = 24; Overall N Lesions PTA = 29
  Participant analysis not performed, as this is a lesion-based measurement.
  mm
    number analyzed (Participants) | 21 | 21 | 42
    number analyzed (Lesions) | 21 | 22 | 43
    (all) | 159.00 (84.66) | 136.43 (72.82) | 147.45 (78.71)
Diameter Stenosis, % [Mean (Standard Deviation); unit: %] — Population: Lesion based measurement. CoreLab reported data; Overall N Lesions DCB = 24; Overall N Lesions PTA = 29
  Participant analysis not performed, as this is a lesion-based measurement.
  %
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 97.59 (6.69) | 96.33 (8.64) | 96.90 (7.77)
Reference vessel diameter, mm [Mean (Standard Deviation); unit: mm] — Population: Lesion based measurement. CoreLab reported data; Overall N Lesions DCB = 24; Overall N Lesions PTA = 29
  Participant analysis not performed, as this is a lesion-based measurement.
  mm
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 2.80 (0.54) | 2.71 (0.39) | 2.75 (0.46)
Minimum lumen diameter, mm [Mean (Standard Deviation); unit: mm] — Population: Lesion based measurement. CoreLab reported data; Overall N Lesions DCB = 24; Overall N Lesions PTA = 29
  Participant analysis not performed, as this is a lesion-based measurement.
  mm
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 0.06 (0.19) | 0.09 (0.21) | 0.08 (0.20)
Calcification [Count of Units; unit: Lesions] — Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 13 | 12 | 25
Calcification - mild/moderate [Count of Units; unit: Lesions] — Calcium is visible along one side of the arterial wall in the area of the target lesion prior to injection of contrast. The calcium present encompasses < 50% of the total target lesion treatment area by visual estimate and/or the calcium is not circumferential (360°) in nature (i.e. on both sides of the vessel lumen extending 2 cm or greater on a single AP view) or classified as exophytic calcification, no impedance of blood flow in the vessel. Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 3 | 4 | 7
Calcification - moderate/severe [Count of Units; unit: Lesions] — Calcium is visible along one or both sides of the arterial wall in the area of the target lesion. The calcium present encompasses ≤ 50% of total target lesion treatment area by visual estimate and/ the calcium is not circumferential (360°) in nature (i.e. on both sides of the vessel lumen extending 2 cm or greater on a single AP view) or classified as exophytic calcification, and does not impede blood flow by more than 50%. Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 8 | 4 | 12
Calcification - severe [Count of Units; unit: Lesions] — Calcium is visible along both sides of the arterial wall, covers 2 cm or greater of the target lesion area, encompasses greater than 50% of the total target lesion treatment area by visual estimate and/or the calcium is circumferential (360°) in nature (i.e. on both sides of the vessel lumen extending 2 cm or greater on a single AP view) or classified as exophytic calcification, significantly impedes blood flow in the vessel. Population: Lesion based measurement. Number of analyzed units corresponds to number of lesions with available data.
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 2 | 4 | 6
TASC II - A [Count of Units; unit: Lesions] — TransAtlantic Inter-Society Consensus; TASC II classification spans from grading A (mildly complex lesions), to D (severe complex lesions). Increased grades indicate more severe lesions. Population: Lesion based measurement. CoreLab reported data; Overall N Lesions DCB = 24; Overall N Lesions PTA = 29
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 1 | 0 | 1
TASC II - B [Count of Units; unit: Lesions] — TransAtlantic Inter-Society Consensus; TASC II classification spans from grading A (mildly complex lesions), to D (severe complex lesions). Increased grades indicate more severe lesions. Population: Lesion based measurement. CoreLab reported data; Overall N Lesions DCB = 24; Overall N Lesions PTA = 29
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 1 | 4 | 5
TASC II - C [Count of Units; unit: Lesions] — TransAtlantic Inter-Society Consensus; TASC II classification spans from grading A (mildly complex lesions), to D (severe complex lesions). Increased grades indicate more severe lesions. Population: Lesion based measurement. CoreLab reported data; Overall N Lesions DCB = 24; Overall N Lesions PTA = 29
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 16 | 17 | 33
TASC II - D [Count of Units; unit: Lesions] — TransAtlantic Inter-Society Consensus; TASC II classification spans from grading A (mildly complex lesions), to D (severe complex lesions). Increased grades indicate more severe lesions. Population: Lesion based measurement. CoreLab reported data; Overall N Lesions DCB = 24; Overall N Lesions PTA = 29
  Participant analysis not performed, as this is a lesion-based measurement.
  Lesions
    number analyzed (Lesions) | 24 | 29 | 53
    (all) | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint: Late Lumen Loss (LLL) at 9 Months
Description: Late lumen loss (LLL) - The difference between minimum lumen diameter (MLD) immediately after percutaneous balloon angioplasty PTA and MLD at follow up, measured at 9 months
Time Frame: 9 Months
Population: 3 participants were missing data in IN.PACT 014 arm, and 3 participants were missing data in the PTA arm.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 20 | 24
mm | 0.892 (0.774) | 1.312 (0.720)

2. Secondary Outcome: Composite Safety Endpoint
Description: A composite of freedom from device- and procedure-related mortality within 30 days, freedom from major target limb amputation and freedom from clinically-driven target lesion revascularization (CD-TLR) within 9 months post-index procedure
Time Frame: 9 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 24
Participants | 21 | 21

3. Secondary Outcome: Major Adverse Event (MAE) Rate
Description: defined as a composite of all-cause mortality, target limb major amputation and clinically-driven target lesion revascularization (CD-TLR)
  Reported by using the event-free survival Kaplan-Meier estimate through 60 months
Time Frame: through 3, 6, 9, 12, 24, 36, 48 and 60 months
Population: number analyzed in one or more rows indicates the number analyzed at each timepoint
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 27
probability
  through 3 months | 95.45 [87.14 to 100] | 96.30 [89.43 to 100]
  through 6 months | 95.45 [87.14 to 100] | 88.89 [77.79 to 100]
  through 9 months | 86.36 [73.15 to 100] | 85.19 [72.79 to 99.70]
  through 12 months | 81.82 [67.19 to 99.63] | 77.78 [63.58 to 95.15]
  through 24 months | 54.55 [37.25 to 79.88] | 70.37 [55.09 to 89.88]
  through 36 months | 45.45 [28.76 to 71.84] | 62.96 [47.15 to 84.09]
  through 48 months | 45.45 [28.76 to 71.84] | 51.16 [35.23 to 74.28]
  through 60 months | 45.45 [28.76 to 71.84] | 46.89 [31.12 to 70.67]

4. Secondary Outcome: Functional Flow Assessment
Description: is defined as absence of target lesion occlusion (no flow) assessed by duplex ultrasound.
Time Frame: at 3, 6, 9, 12, 24 and 36 months
Population: Participant analysis not performed, as this is a lesion-based measurement.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 27
Number analyzed (Lesions) | 24 | 29
Lesions
  At 3 Months: number analyzed (Participants) | 16 | 19
  At 3 Months: number analyzed (Lesions) | 16 | 21
  At 3 Months | 15 | 14
  At 6 Months: number analyzed (Participants) | 17 | 17
  At 6 Months: number analyzed (Lesions) | 17 | 18
  At 6 Months | 15 | 13
  At 9 Months: number analyzed (Participants) | 13 | 10
  At 9 Months: number analyzed (Lesions) | 13 | 10
  At 9 Months | 11 | 6
  At 12 Months: number analyzed (Participants) | 14 | 11
  At 12 Months: number analyzed (Lesions) | 15 | 11
  At 12 Months | 11 | 5
  At 24 Months: number analyzed (Participants) | 8 | 17
  At 24 Months: number analyzed (Lesions) | 8 | 17
  At 24 Months | 6 | 10
  At 36 Months: number analyzed (Participants) | 13 | 13
  At 36 Months: number analyzed (Lesions) | 14 | 15
  At 36 Months | 9 | 6

5. Secondary Outcome: Death of Any Cause
Description: Death of any cause, reported by using the event-free survival Kaplan-Meier estimate through 60 months
Time Frame: through 3, 6, 9, 12, 24, 36, 48 and 60 months
Population: number analyzed in one or more rows indicates the number analyzed at each timepoint
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 27
probability
  Through 3 months | 100.0 [100.0 to 100.0] | 96.30 [89.43 to 100.0]
  Through 6 months | 100.0 [100.0 to 100.0] | 92.59 [83.22 to 100.0]
  Through 9 months | 95.45 [87.14 to 100.0] | 92.59 [83.22 to 100.0]
  Through 12 months | 95.45 [87.14 to 100.0] | 88.89 [77.79 to 100.0]
  Through 24 months | 72.73 [56.31 to 93.94] | 88.89 [77.79 to 100.0]
  Through 36 months | 68.18 [51.25 to 90.71] | 77.78 [63.58 to 95.15]
  Through 48 months | 59.09 [41.74 to 83.66] | 73.89 [58.98 to 92.56]
  Through 60 months | 59.09 [41.74 to 83.66] | 65.68 [49.72 to 86.75]

6. Secondary Outcome: Major Target Limb Amputation Rate
Description: Major Target Limb Amputation rate, reported by using the event-free survival Kaplan-Meier estimate through 60 months
Time Frame: through 30 days, 3, 6, 9, 12, 24, 36, 48 and 60 months
Population: number analyzed in one or more rows indicates the number analyzed at each timepoint
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 27
probability
  Through 30 days | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  Through 3 months | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  Through 6 months | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  Through 9 months | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  Through 12 months | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  Through 24 months | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  Through 36 months | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  Through 48 months | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  Through 60 months | 100.00 [100.00 to 100.00] | 93.75 [82.61 to 100.00]

7. Secondary Outcome: Clinically-driven Target Lesion Revascularization (CD-TLR) Rate
Description: Clinically-driven Target Lesion Revascularization (CD-TLR) rate, reported by using the event-free survival Kaplan-Meier estimate through 60 months
Time Frame: through 3, 6, 9, 12, 24, 36, 48 and 60 months
Population: number analyzed in one or more rows indicates the number analyzed at each timepoint
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 27
probability
  Through 3 months | 95.45 [87.14 to 100.00] | 100.00 [100.00 to 100.00]
  Through 6 months | 95.45 [87.14 to 100.00] | 96.15 [89.04 to 100.00]
  Through 9 months | 90.68 [79.17 to 100.00] | 92.15 [82.27 to 100.00]
  Through 12 months | 85.91 [72.32 to 100.00] | 88.14 [76.39 to 100.00]
  Through 24 months | 80.86 [65.59 to 99.67] | 79.75 [65.34 to 97.33]
  Through 36 months | 73.51 [55.52 to 97.31] | 79.75 [65.34 to 97.33]
  Through 48 months | 73.51 [55.52 to 97.31] | 69.78 [53.16 to 91.60]
  Through 60 months | 73.51 [55.52 to 97.31] | 69.78 [53.16 to 91.60]

8. Secondary Outcome: Mechanically-driven Target Lesion Revascularization (TLR) Rate
Description: Mechanically-driven Target Lesion Revascularization (TLR) rate
Time Frame: through 37 days
Population: Number of subjects undergo MD-TLR within 37 days post-index procedure adjudicated by CEC divided by the number of evaluable subjects at 37 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 26
Participants | 1 | 0

9. Secondary Outcome: Target Lesion Revascularization (TLR) Rate
Description: Target Lesion Revascularization (TLR) rate, reported by using the event-free survival Kaplan-Meier estimate through 60 months
Time Frame: through 3, 6, 9, 12, 24, 36, 48 and 60 months
Population: Number analyzed in one or more rows indicates the number analyzed at each timepoint
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 27
probability
  Through 3 months | 95.65 [87.67 to 100.00] | 100.00 [100.00 to 100.00]
  Through 6 months | 95.65 [87.67 to 100.00] | 96.15 [89.04 to 100.00]
  Through 9 months | 90.87 [79.55 to 100.00] | 84.13 [71.01 to 99.69]
  Through 12 months | 86.09 [72.62 to 100.00] | 80.13 [65.95 to 97.35]
  Through 24 months | 81.02 [65.84 to 99.71] | 71.69 [55.92 to 91.91]
  Through 36 months | 73.66 [55.71 to 97.38] | 71.69 [55.92 to 91.91]
  Through 48 months | 73.66 [55.71 to 97.38] | 62.13 [45.21 to 85.39]
  Through 60 months | 73.66 [55.71 to 97.38] | 62.13 [45.21 to 85.39]

10. Secondary Outcome: Clinically-driven Target Vessel Revascularization (CD-TVR) Rate
Description: Clinically-driven Target Vessel Revascularization (CD-TVR) rate, reported by using the event-free survival Kaplan-Meier estimate through 60 months
Time Frame: through 3, 6, 9, 12, 24, 36, 48 and 60 months
Population: number analyzed in one or more rows indicates the number analyzed at each timepoint
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 27
probability
  Through 3 months | 95.45 [87.14 to 100.00] | 96.15 [89.04 to 100.00]
  Through 6 months | 95.45 [87.14 to 100.00] | 92.31 [82.61 to 100.00]
  Through 9 months | 90.68 [79.17 to 100.00] | 88.29 [76.68 to 100.00]
  Through 12 months | 85.91 [72.32 to 100.00] | 84.28 [71.25 to 99.70]
  Through 24 months | 80.86 [65.59 to 99.67] | 75.85 [60.71 to 94.77]
  Through 36 months | 73.51 [55.52 to 97.31] | 75.85 [60.71 to 94.77]
  Through 48 months | 73.51 [55.52 to 97.31] | 65.74 [48.79 to 88.58]
  Through 60 months | 73.51 [55.52 to 97.31] | 65.74 [48.79 to 88.58]

11. Secondary Outcome: Target Vessel Revascularization (TVR) Rate
Description: Target Vessel Revascularization (TVR) rate, reported by using the event-free survival Kaplan-Meier estimate through 60 months
Time Frame: through 3, 6, 9, 12, 24, 36, 48 and 60 months
Population: number analyzed in one or more rows indicates the number analyzed at each timepoint
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 27
probability
  Through 3 months | 95.65 [87.67 to 100.00] | 96.15 [89.04 to 100.00]
  Through 6 months | 95.65 [87.67 to 100.00] | 92.31 [82.61 to 100.00]
  Through 9 months | 90.87 [79.55 to 100.00] | 80.27 [66.16 to 97.38]
  Through 12 months | 86.09 [72.62 to 100.00] | 76.25 [61.32 to 94.82]
  Through 24 months | 81.02 [65.84 to 99.71] | 67.78 [51.62 to 89.00]
  Through 36 months | 73.66 [55.71 to 97.38] | 67.78 [51.62 to 89.00]
  Through 48 months | 73.66 [55.71 to 97.38] | 58.10 [41.10 to 82.14]
  Through 60 months | 73.66 [55.71 to 97.38] | 58.10 [41.10 to 82.14]

12. Secondary Outcome: Status of Wound Healing
Description: Status of wound healing for baseline wounds: completely healed - improvement - unchanged - worsened - Amputation - skin graft; percentage of wounds in each category is presented for each treatment arm
Time Frame: at 30 days, 3, 6, 9, 12, 24 and 36 months
Population: This is a wound-based measurement. Numbers are % (counts/number of wounds with data).
  Each participant could report one or more baseline wounds, or none. Therefore, the overall number of participants analyzed may not correspond to the number of wounds analyzed. Number of participants analyzed at each timepoint indicates the number of participants with at least one Baseline Wound.
  21 wounds in the IN.PACT 014 arm, and 25 wounds were analyzed in the PTA arm, based on available data.
Measure: Count of Units; unit: Baseline wounds
Units Other Than Participants: Baseline wounds
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 20 | 24
Number analyzed (Baseline wounds) | 21 | 25
Baseline wounds
  Within 30 Days: Completely Healed | 3 | 2
  Within 30 Days: Improvement | 7 | 8
  Within 30 Days: Unchanged | 0 | 3
  Within 30 Days: Worsened | 0 | 1
  Within 30 Days: Amputation | 11 | 11
  Within 30 Days: Skin graft | 0 | 0
  Within 3 Months: number analyzed (Participants) | 20 | 23
  Within 3 Months: number analyzed (Baseline wounds) | 21 | 24
  Within 3 Months: Completely Healed | 5 | 7
  Within 3 Months: Improvement | 4 | 4
  Within 3 Months: Unchanged | 0 | 2
  Within 3 Months: Worsened | 1 | 0
  Within 3 Months: Amputation | 11 | 11
  Within 3 Months: Skin graft | 0 | 0
  Within 6 Months: number analyzed (Participants) | 20 | 23
  Within 6 Months: number analyzed (Baseline wounds) | 21 | 24
  Within 6 Months: Completely Healed | 8 | 10
  Within 6 Months: Improvement | 2 | 0
  Within 6 Months: Unchanged | 0 | 1
  Within 6 Months: Worsened | 0 | 1
  Within 6 Months: Amputation | 11 | 12
  Within 6 Months: Skin graft | 0 | 0
  Within 9 Months: number analyzed (Participants) | 20 | 22
  Within 9 Months: number analyzed (Baseline wounds) | 21 | 23
  Within 9 Months: Completely Healed | 9 | 10
  Within 9 Months: Improvement | 1 | 1
  Within 9 Months: Unchanged | 0 | 1
  Within 9 Months: Worsened | 0 | 0
  Within 9 Months: Amputation | 11 | 11
  Within 9 Months: Skin graft | 0 | 0
  Within 12 Months: number analyzed (Participants) | 19 | 22
  Within 12 Months: number analyzed (Baseline wounds) | 20 | 23
  Within 12 Months: Completely Healed | 8 | 10
  Within 12 Months: Improvement | 1 | 0
  Within 12 Months: Unchanged | 0 | 2
  Within 12 Months: Worsened | 0 | 0
  Within 12 Months: Amputation | 11 | 11
  Within 12 Months: Skin graft | 0 | 0
  Within 24 Months: number analyzed (Participants) | 19 | 21
  Within 24 Months: number analyzed (Baseline wounds) | 20 | 22
  Within 24 Months: Completely Healed | 8 | 9
  Within 24 Months: Improvement | 1 | 0
  Within 24 Months: Unchanged | 0 | 2
  Within 24 Months: Worsened | 0 | 0
  Within 24 Months: Amputation | 11 | 11
  Within 24 Months: Skin graft | 0 | 0
  Within 36 Months: number analyzed (Participants) | 13 | 21
  Within 36 Months: number analyzed (Baseline wounds) | 13 | 22
  Within 36 Months: Completely Healed | 6 | 9
  Within 36 Months: Improvement | 0 | 0
  Within 36 Months: Unchanged | 0 | 2
  Within 36 Months: Worsened | 0 | 0
  Within 36 Months: Amputation | 7 | 11
  Within 36 Months: Skin graft | 0 | 0

13. Secondary Outcome: Rate of Thrombosis at the Target Lesion
Description: Rate of thrombosis at the target lesion, reported by using the event-free survival Kaplan-Meier estimate through 60 months
Time Frame: through 30 days, 3, 6, 9, 12, 24, 36, 48 and 60 months
Population: number analyzed in one or more rows indicates the number analyzed at each timepoint
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 27
probability
  Through 30 days | 95.7 [87.6 to 100.0] | 96.3 [89.4 to 100.0]
  Through 3 months | 95.7 [87.6 to 100.0] | 96.3 [89.4 to 100.0]
  Through 6 months | 95.7 [87.6 to 100.0] | 96.3 [89.4 to 100.0]
  Through 9 months | 95.7 [87.6 to 100.0] | 96.3 [89.4 to 100.0]
  Through 12 months | 90.9 [79.5 to 100.0] | 96.3 [89.4 to 100.0]
  Through 24 months | 86.1 [72.6 to 100.0] | 96.3 [89.4 to 100.0]
  Through 36 months | 86.1 [72.6 to 100.0] | 96.3 [89.4 to 100.0]
  Through 48 months | 86.1 [72.6 to 100.0] | 96.3 [89.4 to 100.0]
  Through 60 months | 86.1 [72.6 to 100.0] | 96.3 [89.4 to 100.0]

14. Secondary Outcome: Device Success
Description: Calculated as the number of IN.PACT 014 Investigational devices with successful delivery, balloon inflation, deflation and retrieval of the intact study device without burst below the rated burst pressure (RBP), divided by the total number of IN.PACT 014 Investigational devices assessed in the study
Time Frame: at the time of procedure
Population: 68 IN.PACT 014 Investigational devices used
Measure: Count of Units; unit: IN.PACT 014 Investigational devices
Units Other Than Participants: IN.PACT 014 Investigational devices
Arm/Group | Drug Coated Balloon IN.PACT 014
Number analyzed (Participants) | 23
Number analyzed (IN.PACT 014 Investigational devices) | 68
IN.PACT 014 Investigational devices | 64

15. Secondary Outcome: Clinical Success
Description: Clinical success is defined as residual stenosis of ≤ 30% without procedural complications (death, major target limb amputation, thrombosis of the target lesion, or target vessel revascularization (TVR)). If any lesion has residual stenosis > 30% or any of the complications (death, major target limb amputation, thrombosis of the target lesion, or TVR) prior to discharge, then subject is not counted as having Clinical Success.
  Clinical success is calculated as the number of index procedures with residual stenosis of ≤ 30% by core lab (use site reported data if core lab data is not available) for all target lesions and without procedural complications (death, major target limb amputation, thrombosis of the target lesion, or TVR) prior to discharge as adjudicated by CEC, divided by the number of total index procedures performed.
Time Frame: up to discharge visit [between index procedure and 30-day (+/- 7 days) follow-up visit. The average days until discharge was: 9 days (with a max. of 31days) in the IN.PACT 014 arm, and 6 days (with a max. of 21days) in the PTA arm.]
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
Number analyzed (Participants) | 23 | 27
Participants | 12 | 11

ADVERSE EVENTS:
Time Frame: 1800 Days (60 Months)
Arm/Group | Drug Coated Balloon IN.PACT 014 | Percutaneous Transluminal Angioplasty (PTA)
All-Cause Mortality (participants affected / at risk) | 9/23 | 9/27
Serious Adverse Events (participants affected / at risk) | 19/23 | 25/27
Other Adverse Events (participants affected / at risk) | 13/23 | 24/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug Coated Balloon IN.PACT 014 (N=23) | Percutaneous Transluminal Angioplasty (PTA) (N=27)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 1
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 1
CARDIAC FAILURE (Cardiac disorders) | 5 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 | 3
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 | 1
MICROVASCULAR CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 2
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 1 | 0
FOOD POISONING (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 2 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0
DEATH (General disorders) | 1 | 1
IMPAIRED HEALING (General disorders) | 0 | 1
VASCULAR STENT OCCLUSION (General disorders) | 0 | 1
VASCULAR STENT THROMBOSIS (General disorders) | 1 | 1
BILE DUCT STONE (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 2
COVID-19 PNEUMONIA (Infections and infestations) | 1 | 1
ENDOCARDITIS (Infections and infestations) | 0 | 1
ENDOCARDITIS PSEUDOMONAL (Infections and infestations) | 1 | 0
GANGRENE (Infections and infestations) | 1 | 3
INFECTED SKIN ULCER (Infections and infestations) | 0 | 1
KLEBSIELLA INFECTION (Infections and infestations) | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 | 3
SEPSIS (Infections and infestations) | 1 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 1
UROSEPSIS (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 2 | 3
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 2 | 4
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
PERIPHERAL ARTERIAL REOCCLUSION (Injury, poisoning and procedural complications) | 3 | 8
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 3 | 4
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 3 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
METASTATIC GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 | 0
SPONDYLITIC MYELOPATHY (Nervous system disorders) | 0 | 1
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 1 | 0
DEVICE DEFECTIVE (Product Issues) | 1 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 2
HAEMATURIA (Renal and urinary disorders) | 0 | 1
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2
DIABETIC WOUND (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 1
ISCHAEMIC SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 6
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 3 | 2
CARDIAC PACEMAKER REPLACEMENT (Surgical and medical procedures) | 0 | 1
PERIPHERAL ARTERY ANGIOPLASTY (Surgical and medical procedures) | 0 | 1
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 1 | 0
EXTREMITY NECROSIS (Vascular disorders) | 1 | 1
ISCHAEMIA (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 2
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 5 | 8
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 2 | 4
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 4 | 2
PERIPHERAL ISCHAEMIA (Vascular disorders) | 3 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drug Coated Balloon IN.PACT 014 (N=23) | Percutaneous Transluminal Angioplasty (PTA) (N=27)
IMPAIRED HEALING (General disorders) | 1 | 2
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 4
PERIPHERAL ARTERIAL REOCCLUSION (Injury, poisoning and procedural complications) | 2 | 6
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 2 | 5
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 3
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 2 | 0
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 2 | 0
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 2 | 3
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT02963649/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT02963649/SAP_001.pdf